CLINICAL TRIAL: NCT02673216
Title: Infection and Adverse Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Statens Serum Institut (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-116-14
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Vaginal Swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spontaneous abortion: Women attending for suspected spontaneous abortion
  Interventions: Other: No intervention
- Normal pregnant women: Normal pregnant women attending for nuchal translucency scan
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Miscarriage (spontaneous abortion, stillbirth, and preterm birth) is the most common adverse out-come of pregnancy and a significant proportion is caused by infection. The investigators aim to study vaginal specimens from 1200 pregnant women recruited before 14 weeks of gestation with follow-up at mid-term (week 19) as well as 300 women aborting spontaneously. Adverse pregnancy outcome will be correlated to the presence of bacterial vaginosis (BV) subclasses, to vaginal fluid inflammation markers, and to the presence of novel Chlamydia-like bacteria, in particular Waddlia chondrophila. Species specific quantitative PCR assays for BV-related bacteria as well as next-generation-sequencing will be applied on selected specimens with the aim to identify markers allowing for a personalised treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending for antenatal care or with spontaneous miscarriage
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Preterm birth <37 weeks of gestation | 37 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen S Jensen, DMedSci, PhD, Principal Investigator — Statens Serum Institut
Locations (1):
- Skejby University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No